CLINICAL TRIAL: NCT02341521
Title: An Evaluation of the Plasma and Urine Pharmacokinetics of Parent Compound and a Metabolite of OC000459 in Healthy Male and Female Subjects
Brief Title: Evaluation of Metabolic Profile of OC000459
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atopix Therapeutics, Ltd. (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OC000459/018/14
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OC000459 50 mg (Experimental): OC000459 50 mg daily for 8 days
  Interventions: Drug: OC000459

INTERVENTIONS:
Drug: OC000459 — Taken orally for 8 days

SUMMARY:
An open label study in 9 male and 9 female healthy subjects to determine the pharmacokinetics of parent compound and metabolite after eight days of dosing.

DETAILED DESCRIPTION:
The study will include 9 male and 9 female healthy subjects. Following informed consent and satisfactory screening, each will be dosed for seven consecutive days on an outpatient basis with OC000459 50 mg daily taken before breakfast. On the seventh day, subjects will report to the clinical unit. Following an overnight fast, blood samples will be drawn for baseline safety and pharmacokinetic measurements and a urine specimen will be obtained for urinalysis and baseline metabolite measurements and subjects will be dosed with 50 mg OC000459. Blood samples will then be drawn at selected intervals for 120 hours post dosing and will be analysed for OC000459 parent compound and its metabolite. Urine collections will be obtained over the same period to determine the excretion of the metabolite and parent compound in urine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, any racial group
2. Aged 18-55 years inclusive
3. Able to comply with the protocol
4. Subjects with a Body Mass Index (BMI) of 21-28 (BMI = Body weight (kg) / (Height (m)2)
5. Subjects with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 21 days of the first dose

Exclusion Criteria:

1. A history of gastrointestinal disorder likely to influence drug absorption
2. Receipt of any medication including over the counter preparations and vitamins within 14 days of the first study day with the exception of paracetamol up to a maximum of 2 g daily
3. Evidence of clinically significant renal, hepatic, cardiovascular or metabolic dysfunction
4. A history of drug or alcohol abuse
5. Inability to communicate well with the investigator (i.e., language problem, poor mental development or impaired cerebral function)
6. Participation in a clinical study within 3 months of the first dose of study drug. Subjects will be checked against The Over Volunteering Prevention System (TOPS)
7. Donation of 450 mL or more blood within 60 days of the first dose of study drug
8. A history of hypersensitivity and/or idiosyncrasy to any of the test compounds or related drugs or excipients employed in this study
9. Pregnancy or lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Metabolite | Day 8
  Metabolite AUC

SECONDARY OUTCOMES:
Parent compound | Day 8
  Parent compound AUC

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Merthyr Tydfil, Wales, United Kingdom